CLINICAL TRIAL: NCT06750393
Title: Combined Effects of Barre and Gym Ball Exercises on Pain, Distress and Quality of Life in Primary Dysmenorrhoea
Brief Title: Combined Effects of Barre and Gym Ball Exercises in Primary Dysmenorhoea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0528
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Dysmenorrhea Primary
Keywords: gym; exercises; quality of life; dysmenorrhea; Menstrual Cycle; female
MeSH Terms: conditions — Motor Activity; Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barre exercise with gym ball exercise (Experimental): The Barre exercises will be administered to the participant of Group A for a period of 3 month. Each exercise will be given for 10 s hold × 12 times/set × 3 sets/day × 3 days/week
  × 12. Gym ball exercises program include Knee tucks, leg curls, back extension exercises
  Interventions: Other: Barre exercise along with gym ball exercises
- Barre exercises (Active Comparator): The Barre exercises for a period of 3 month Each exercise will be given for 10 s hold × 12 times/set × 3 sets/day × 3 days/week
  × 12. During
  Interventions: Other: Barre exercises

INTERVENTIONS:
Other: Barre exercise along with gym ball exercises — The Barre exercises will be administer to the participant of Group A for a period of 3 month.
  Each exercise will be given for 10 s hold × 12 times/set × 3 sets/day × 3 days/week
  × 12. Gym ball exercises program include Knee tucks, leg curls, back extension exercises
  Arms: Barre exercise with gym ball exercise
Other: Barre exercises — The Barre exercises for a period of 3 month Each exercise will be given for 10 s hold × 12 times/set × 3 sets/day × 3 days/week
  × 12. During
  Arms: Barre exercises

SUMMARY:
Group A will be given Barre and gym ball exercises. Group B will be given Barre exercises. All these sessions will be of 30-minute 3session per week for 12 weeks.

DETAILED DESCRIPTION:
This will be a randomized controlled trial conducted on 42 participants. Data will be collected from USKT (University of Sialkot) and UMT (University of Management and Technology Sialkot by using non-probability convenience sampling technique. WaLLiD score scale is used to determine the severity of dysmenorrhoea. Girls between the age of 17 to 25 with history of dysmenorrhea will be included in this study. Participants who has history of secondary dysmenorrhea, Diagnosed with polycystic ovarian syndrome will be excluded from this study. A sample of 42 will be divided in to two groups with 21 participants in each group. Group A will be given Barre and gym ball exercises. Group B will be given Barre exercises. All these sessions will be of 30 minute 3session per week for 12 weeks. Pre and post assessment of pain, distress , severity of dysmenorrhoea and quality of life will be done by using numeric pain rating scale, menstrual distress questionnaire, WaLLiD scale and Q-LES-Q-SF questionnaire. Data will be analyzed by using SPSS version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Female suffered from primary dysmenorrhea diagnosed through WaLLiD score range from 5-12
* Female having 5 and above score on Numerical Pain Rating Scale
* Female having regular menstrual period form at least 3 months
* Female having a history of dysmenorrhea occurring at least three times in the past six months

Exclusion Criteria:

* Females using hormonal contraception.
* Females who are married.
* Females with secondary dysmenorrhea
* Females diagnosed with polycystic ovarian syndrome
* Females having menstrual issues
* Females who take analgesic
* Females having BMI > 25
* Participants who show unwillingness to participate in the study

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — diagnosed with primary dysmenorrhea
Enrollment: 42 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain rating Scale | 12th week
  Numeric pain rating scale is a subjective measure 11 point numerical scale which is used to measure pain. Is scoring range In this scale 0 shows no pain and 10 shows worst pain imaginable. It has good reliability of 0.79 and validity of 0.96.
Menstrual distress questionnaire (MEDI-Q): | 12th week
  The Menstrual Distress Questionnaire (MEDI-Q) is a newly developed tool that has been validated for comprehensive evaluation of menstrual-related distress .It consists of 25 items that cover different areas of menstruation-related symptoms, such as pain, discomfort, psychic or cognitive changes, and gastrointestinal disturbances. In this scale 0 -16 score indicates Mild symptoms, indicating minimal distress,17-34 indicates Moderate symptoms, indicating moderate distress.35-56 indicates Severe symptoms. It is reliable tool with reliability 0.84 and validity 0.95.
Quality Of Life Enjoyment And Satisfaction Questionnaire Short Form(Q-LESQ-SF) | 12th week
  Short-Form (Q-LES-Q-SF) was derived from the general activities scale of the original 93- item questionnaire. It consists of 16 items but only 14 item scores are computed, the last two are stand-alone items. Q-LES-Q-SF is rated on a 5-point scale as 1-very poor, 2-poor, 3-fair, 4-good, and 5-very good. 70 is the maximum score. It is a reliable and valid tool with values 0.9 and 0.93.
WaLLiD Score | 12th week
  WaLLiD score was designed to diagnose dysmenorrhea and predict medical leave score as a standard survey that validated and constructed the classification of the severity of dysmenorrhea. The interpretation of the WaLLiD questionnaire is as follows: 0 = No dysmenorrhea 1-4 =Mild dysmenorrhea 5-7 = Moderate dysmenorrhea 8-12 = Severe dysmenorrhea WaLLiD score is reliable tool with value of 0.723

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- University of Sialkot, University of Management Technology, Sialkot, Pjunjab, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samperio MM, Pardo ACJMSR. Efectos del ejercicio físico en la dismenorrea primaria. Revisión sistemática. 2021;1(1).
- [Background] Azabu A, Fernandes P, Thomas T. Effect Of a Gym Ball Exercise Program on Dysmenorrhea in Nursing Students of a Selected College in Mangaluru, India: A Quasi experimental Study. gums-hnmj. 2024;34(1):29-34
- [Background] Lopez-Liria R, Torres-Alamo L, Vega-Ramirez FA, Garcia-Luengo AV, Aguilar-Parra JM, Trigueros-Ramos R, Rocamora-Perez P. Efficacy of Physiotherapy Treatment in Primary Dysmenorrhea: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jul 23;18(15):7832. doi: 10.3390/ijerph18157832. PMID 34360122
- [Background] .Krasova I, Semyzorova A, Deineko A, Beihul I, Shyshkina OJPR, Technologies RH. Barre fitness as a modern means of improving the health of women in the first period of adulthood. 2023;8(1):29-38
- [Background] Hidayah N, Fatmawati R. The effectiveness of Gym Ball and ambon banana consumption against menstrual pain reduction in teenagers. 2022.
- [Background] Hemalatha R, Shanmugananth E, Murugaraj T, Velkumar VJJoCLM. Effects of Barre Exercise Versus Pilates Versus Aerobic Exercise on Pre-Menstrual Syndrome Among College Going Coastal Students. 2023;11:2440-51.
- [Background] Tianing NW, Nugraha MHS, Indrayani AW, Widyadharma IPEJBMJ. The difference in the effectiveness of warm compress and active stretching exercise in reducing dysmenorrhea pain. 2021;10(3):1041-4.
- [Background] Ali Z, Cardoza J. A Study on Effects of Aerobic Exercises on Quality of Life in Primary Dysmenorrhea in Bangalore. Natural Volatiles and Essential Oils. 2021;8:5304-12.